CLINICAL TRIAL: NCT04930913
Title: The Value of Three-dimensional Ultrasound Applying in Pre and Postoperative Assessment and Prognosis of Intrauterine Adhesions
Brief Title: Three-dimensional Ultrasound Applying in Assessment of Intrauterine Adhesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Xiaowu Huang, Director of department, Fu Xing Hospital, Capital Medical University
Other Study IDs: 2020-1-7027
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Three-dimensional Ultrasound — women suspected of having adhesions will perform 3D US

SUMMARY:
In this prospective, multicenter, large-scale study，the investigators wish to examine the accuracy of several three-dimensional ultrasound anatomical and vascular parameters in diagnosing IUA when compared to the gold standard of hysteroscopy，and to assess the value of 3D US applying in prognosis of intrauterine adhesions.

DETAILED DESCRIPTION:
1. Study Design This is a prospective, multicenter, large-scale diagnostic testing. We use hysteroscopy finding as standard reference.
2. Study population 600 patients from three tertiary hospitals suspected of having IUA will be prospectively recruited. Thorough assessment including previous reproductive and surgical history as well as menstrual pattern will be performed.
3. Study Procedure 3.1 Diagnosis

IUA will be diagnosed in coronal plane, based on a suggestion reported by a Taiwanese study. The morphological characteristics of the endometrium suggesting IUA include as follow:

* marginal irregularity (in coronal plane)
* defects (interrupted endometrial line)
* obliteration (undetectable endometrium suggesting extensive adhesion)
* fibrosis or calcification (hyperechoic lesion without posterior shadowing, or with posterior shadowing) 3.2 Ultrasound
* Transvaginal Ultrasound will be performed in luteal phase.
* Using E10 Voluson GE with 3D/4D TV probe.
* Scan and rendering will be performed in a standardized technique (omniview mode).
* Several parameters will be measured including endometrial volume, uterine volume, vascularization (VI FI VFI).

3.3 Hysteroscopy

* Hysteroscopic exam will be used as the gold standard for the diagnosis of intrauterine adhesions.
* hysteroscopy will confirm the presence, extent, and morphological characteristics of adhesions and the quality of the endometrium.

3.4 Surgical technique

* Hysteroscopic surgery will be performed in a standardized manner.
* The severity and extent of intrauterine adhesions will be scored according to different classification systems. (ESGE/AFS/China consensus)
* a Foley-catheter filled with 3.0ml normal saline will be inserted into the uterus for 5-7 days after surgery.

3.5 Postoperative treatments

* All subjects will be treated with Hormone therapy for at least 8 weeks
* A second-look hysteroscopy will be carried out 4 weeks after surgery, a third-look hysteroscopy will be carried out 12 weeks after surgery
* A second-look 3D US will be carried out in luteal phase after two menstrual peroid postoperatively.

3.6 Follow up

* Follow-up styles: the doctor's outpatient review, telephone, WeChat and so on.
* Follow-up time:3 months, 6months, 12 months after the operation.
* Follow up the results of hysteroscopy and 3D US at 3 months after the operation and the menstrual improvement at 6months after the operation and pregnancy outcomes at 12 months after the operation

ELIGIBILITY:
Inclusion Criteria:

* women aged 20-40
* oligomenorrhea or amenorrhea
* BMI 18-30
* regular menstruation
* written consent obtained

Exclusion Criteria:

* Hypothalamic amenorrhea, pituitary amenorrhea and ovarian amenorrhea
* Patients with uterine fibroids, adenomyosis, uterine malformation and endometrial polyps
* Patients with uterine artery embolization
* History of endometrial hyperplasia
* Irregular menstruation
* Patients with severe complications
* Patients with hypoovarian function

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 600 patients from three Tertiary hospitals suspected of having IUA will be prospectively recruited
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Endometrial volume | 1 year
  Endometrial volume will be measured in in luteal phase by 3D US

CONTACTS AND LOCATIONS:
Overall Officials: Li Tinchiu, Study Chair — Fuxing Hospital,Capital Medical University
Locations (1):
- Fu Xing Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim MJ, Lee Y, Lee C, Chun S, Kim A, Kim HY, Lee JY. Accuracy of three dimensional ultrasound and treatment outcomes of intrauterine adhesion in infertile women. Taiwan J Obstet Gynecol. 2015 Dec;54(6):737-41. doi: 10.1016/j.tjog.2015.10.011. PMID 26700995
- [Background] Amin TN, Saridogan E, Jurkovic D. Ultrasound and intrauterine adhesions: a novel structured approach to diagnosis and management. Ultrasound Obstet Gynecol. 2015 Aug;46(2):131-9. doi: 10.1002/uog.14927. Epub 2015 Jul 20. No abstract available. PMID 26094824
- [Background] Carrascosa P, Capunay C, Vallejos J, Carpio J, Baronio M, Papier S. Two-dimensional and three-dimensional imaging of uterus and fallopian tubes in female infertility. Fertil Steril. 2016 Jun;105(6):1403-1420.e7. doi: 10.1016/j.fertnstert.2016.04.016. Epub 2016 Apr 29. PMID 27140290
- [Background] AAGL Elevating Gynecologic Surgery. AAGL practice report: practice guidelines on intrauterine adhesions developed in collaboration with the European Society of Gynaecological Endoscopy (ESGE). Gynecol Surg. 2017;14(1):6. doi: 10.1186/s10397-017-1007-3. Epub 2017 May 1. No abstract available. PMID 28603474
- [Background] Salazar CA, Isaacson K, Morris S. A comprehensive review of Asherman's syndrome: causes, symptoms and treatment options. Curr Opin Obstet Gynecol. 2017 Aug;29(4):249-256. doi: 10.1097/GCO.0000000000000378. PMID 28582327
- [Background] Dreisler E, Kjer JJ. Asherman's syndrome: current perspectives on diagnosis and management. Int J Womens Health. 2019 Mar 20;11:191-198. doi: 10.2147/IJWH.S165474. eCollection 2019. PMID 30936754